CLINICAL TRIAL: NCT01996332
Title: An Open-label Study of the Effect of Tarceva Monotherapy on Treatment Response in Patients With Advanced Non-small Cell Lung Cancer for Whom Tarceva Monotherapy is Considered the Best Option
Brief Title: A Study of Tarceva (Erlotinib) Monotherapy in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML17915
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Results first posted 2014-07-10 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-06

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

ARMS (1):
- Tarceva Arm (Experimental)
  Interventions: Drug: erlotinib [Tarceva]

INTERVENTIONS:
Drug: erlotinib [Tarceva] — 150 mg/day until progressive disease or unacceptable toxicity

SUMMARY:
This study will evaluate the efficacy and safety of oral Tarceva in patients with advanced NSCLC for whom Tarceva monotherapy is considered the best therapeutic option. The anticipated time on study treatment is 3-12 months.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >=18 years of age;
* locally advanced or metastatic NSCLC (Stage IIIB or IV);
* not a candidate for curative surgery or radical chemotherapy;
* no brain metastases, or clinically stable metastases for >=2 months.

Exclusion Criteria:

* radiotherapy over the previous 2 weeks;
* weight loss >10% in the previous 6 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1805 (Actual)
Dates: Start 2004-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (63):
- Spain (63):
  - Alcoy, Alicante
  - Alicante, Alicante
  - Elche, Alicante
  - Almería, Almeria
  - Ávila, Avila
  - Badajoz, Badajoz
  - Don Benito, Badajoz
  - Mérida, Badajoz
  - Ibiza Town, Balearic Islands
  - Palma de Mallorca, Balearic Islands
  - Badalona, Barcelona
  - Barcelona, Barcelona
  - Granollers, Barcelona
  - Manresa, Barcelona
  - Mataró, Barcelona
  - Sabadell, Barcelona, Barcelona
  - Sant Coloma Gramenet, Barcelona
  - Sant Pere de Ribes, Barcelona
  - Terrassa, Barcelona
  - Vic, Barcelona
  - Burgos, Burgos
  - Cáceres, Caceres
  - Algeciras, Cadiz
  - Cadiz, Cadiz
  - Jerez de la Frontera, Cadiz
  - Puerto Real, Cadiz
  - Santander, Cantabria
  - Torrevieja, Cantabria
  - Castellon, Castellon
  - Córdoba, Cordoba
  - Girona, Girona
  - Baza, Granada
  - Granada, Granada
  - Donostia / San Sebastian, Guipuzcoa
  - Huelva, Huelva
  - Jaén, Jaen
  - A Coruña, La Coruña
  - Ferrol, La Coruña
  - Las Palmas de Gran Canaria, Las Palmas
  - León, Leon
  - Lleida, Lerida
  - Lugo, Lugo
  - Alcorcón, Madrid
  - Madrid, Madrid
  - Málaga, Malaga
  - Cartagena, Murcia
  - Murcia, Murcia
  - Navarra, Navarre
  - Pamplona, Navarre
  - Ourense, Orense
  - Palencia, Palencia
  - Vigo, Pontevedra
  - Salamanca, Salamanca
  - Segovia, Segovia
  - Seville, Sevilla
  - San Cristóbal de La Laguna, Tenerife
  - Santa Cruz de Tenerife, Tenerife
  - Sagunto, Valencia
  - Valencia, Valencia
  - Valladolid, Valladolid
  - Barakaldo, Vizcaya
  - Bilbao, Vizcaya
  - Zaragoza, Zaragoza

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three cohorts were established in participants with advanced non-small cell lung cancer (NSCLC) based on previous chemotherapy treatment received: first line of treatment (where conventional chemotherapy is not indicated), second line of treatment, and third and subsequent lines of treatment. Inclusion was competitive.
Groups:
- Erlotinib 150 Milligrams Per Day (mg/Day): Participants received erlotinib 150 milligrams/day (mg/day), orally, until progressive disease or unacceptable toxicity.
Period: Overall Study
Arm/Group | Erlotinib 150 Milligrams Per Day (mg/Day)
Started | 1805
Completed | 0
Not Completed | 1805
Not completed — Adverse Event | 117
Not completed — Lack of Efficacy | 1245
Not completed — Death | 264
Not completed — Protocol Violation | 9
Not completed — Withdrawal by Subject | 71
Not completed — Other | 20
Not completed — Clinical Deterioration | 28
Not completed — Physician Decision | 17
Not completed — Lost to Follow-up | 34

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population defined as all participants included to each of three cohorts based on prior chemotherapy treatment received: first-line monotherapy (for whom conventional chemotherapy was not indicated), second-line monotherapy, and third or subsequent lines of treatment.
Groups:
- Erlotinib 150 mg/Day: Participants received erlotinib 150 mg/day, orally, until progressive disease or unacceptable toxicity.
Arm/Group | Erlotinib 150 mg/Day
Number analyzed (Participants) | 1805
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.55 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 520
  Male | 1285

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression or Death by Line of Treatment
Description: Time to progression or death was defined as the time from inclusion to the date of disease progression or death, whichever occurred first.
Time Frame: Baseline, every 6-8 weeks up to 3 years until disease progression or death
Population: ITT Population; data were analyzed in 6 cohorts, with erlotinib treatment as: 1) first line; 2) maintenance after first line; 3) second line; 4) maintenance after second line; 5) third or subsequent line; or 6) maintenance after third line
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib 150 mg/Day
Number analyzed (Participants) | 1805
months
  1st Line | 3.4 [2.9 to 4.1]
  Maintenance after 1st Line | 4.7 [3.0 to 6.6]
  2nd Line | 2.7 [2.5 to 2.9]
  Maintenance after 2nd Line | 3.9 [1.2 to 6.8]
  3rd or Subsequent Line | 2.4 [2.2 to 2.7]
  Maintenance after 3rd Line | 2.8 [1.8 to 5.0]

2. Secondary Outcome: Percentage of Participants Achieving Clinical Benefit by Line of Treatment
Description: Efficacy was analyzed in terms of clinical benefit, defined as the sum of the number of participants achieving complete response [CR], partial response [PR], or stable disease [SD]. Tumor response was evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.0. CR was defined as disappearance of all target and non-target lesions. PR was defined as greater than or equal to (≥)30 percent (%) decrease in sum of longest diameters of target lesions taking as reference baseline sum longest diameters associated to non-progressive disease response for non target lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease taking as reference smallest sum of longest dimensions since treatment started associated to non-progressive disease response for non target lesions.
Time Frame: Baseline, every 6-8 weeks up to 3 years or until death
Population: Response evaluable population: participants with measurable disease and with matching criteria to have a response assessment; data were analyzed in 6 cohorts, with erlotinib treatment as: 1) first line; 2) maintenance after first line; 3) second line; 4) maintenance after second line; 5) third or subsequent line; or 6) maintenance after third line
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib 150 mg/Day
Number analyzed (Participants) | 1261
percentage of participants
  1st line | 70.32 [65.21 to 75.08]
  Maintenance treatment after 1st line | 70.00 [53.47 to 83.44]
  2nd line | 58.04 [53.39 to 62.60]
  Maintenance treatment after 2nd line | 73.68 [48.80 to 90.85]
  3rd or subsequent line | 52.71 [47.61 to 57.78]
  Maintenance treatment after 3rd line | 50.00 [15.70 to 84.30]

3. Secondary Outcome: Overall Survival (OS) by Line of Treatment
Description: Time in months from the start of study treatment to date of death due to any cause. OS was calculated as (the death date or last known alive date [if death date was unavailable] minus the date of first dose of study medication plus 1 divided by 30.44).
Time Frame: Baseline, every 6-8 weeks up to 3 years, or until death
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib 150 mg/Day
Number analyzed (Participants) | 1805
months
  1st Line | 6.4 [5.8 to 7.4]
  Sequential treatment after 1st line | 12.1 [6.2 to 19.3]
  2nd Line | 5.9 [5.2 to 6.4]
  Sequential treatment after 2nd line | 7.1 [2.2 to 15.8]
  3rd Line or subsequent | 5.2 [4.3 to 6.1]
  Sequential treatment after 3rd line | 3.9 [2.0 to 8.6]

ADVERSE EVENTS:
Time Frame: From the administration of first dose of study medication to the end of study or until death.
Description: Nonserious adverse events presented in this record include all adverse events reported during the study, not just nonserious events.
Arm/Group | Erlotinib 150 mg/Day
Serious Adverse Events (participants affected / at risk) | 566/1805
Other Adverse Events (participants affected / at risk) | 1695/1797
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib 150 mg/Day (N=1805)
Hemoglobbin (Blood and lymphatic system disorders) | 3
Neutrophils (Investigations) | 2
Platelets (Investigations) | 1
Cardiac arrhythmia (Cardiac disorders) | 4
Cardiac ischemia (Cardiac disorders) | 6
Cardiopulmonary arrest (Cardiac disorders) | 6
Hypotension (Vascular disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 4
Pericardial effusion (Cardiac disorders) | 7
Pericarditis (Cardiac disorders) | 1
Right ventricular dysfunction (Cardiac disorders) | 1
Alcohol Poisoning (Injury, poisoning and procedural complications) | 1
Asthenia (General disorders) | 17
Constitutional symptoms/other (General disorders) | 14
Drug abuser (Social circumstances) | 1
Fever (General disorders) | 17
Opioid abuse (Social circumstances) | 2
Sweating (Skin and subcutaneous tissue disorders) | 1
Weight loss (Investigations) | 1
Dermatology/skin - other (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 6
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 28
Dyspepsia/heartburn (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 6
Esophagitis (Gastrointestinal disorders) | 1
Gastrointestinal/other (Gastrointestinal disorders) | 1
Ileus GI (Gastrointestinal disorders) | 4
Intestinal perforation (Gastrointestinal disorders) | 2
Mucositis (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 6
Obstruction/GU (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 21
Hemorrhage (Blood and lymphatic system disorders) | 17
Hepatic cyst (Hepatobiliary disorders) | 1
Liver dysfunction (Hepatobiliary disorders) | 4
Febrile neutropenia (Infections and infestations) | 2
Gallbladder infection (Infections and infestations) | 1
Infection NOS (Infections and infestations) | 67
Infection - anal/perianal (Infections and infestations) | 1
Infection - appendix (Infections and infestations) | 1
Infection - blood (Infections and infestations) | 6
Infection - brain (encephalitis, infectious) (Infections and infestations) | 1
Infection - bronchus (Infections and infestations) | 5
Infection - catheter - related (Infections and infestations) | 1
Infection - kidney (Infections and infestations) | 1
Infection - liver (Infections and infestations) | 1
Infection - lung (pneumonia) (Infections and infestations) | 44
Infection - skin (cellulitis) (Infections and infestations) | 2
Infection - soft tissue NOS (Infections and infestations) | 3
Infection - upper aerodigestive NOS (Infections and infestations) | 1
Infection - urinary tract NOS (Infections and infestations) | 6
Infection - wound (Infections and infestations) | 1
Edema Limb (General disorders) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Bilirubin (Investigations) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 1
Ascites (Gastrointestinal disorders) | 2
Fracture (Injury, poisoning and procedural complications) | 4
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/other (Musculoskeletal and connective tissue disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 2
CNS ischemia (Nervous system disorders) | 14
Cognitive disturbance (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 11
Dizziness (Nervous system disorders) | 3
Encephalopathy (Nervous system disorders) | 1
Involuntary movement (Nervous system disorders) | 1
Mood alteration - agitation (Psychiatric disorders) | 2
Mood alteration - anxiety (Psychiatric disorders) | 2
Neurology/other (Psychiatric disorders) | 15
Neuropathy/motor (Nervous system disorders) | 7
Neuropathy/sensory (Nervous system disorders) | 2
Psychosis (Psychiatric disorders) | 1
Seizures (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 2
Speech impairment (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 4
Diplopia (Eye disorders) | 1
Keratitis (Eye disorders) | 1
Pain NOS (General disorders) | 22
Pain - abdominal NOS (Gastrointestinal disorders) | 7
Pain - bone (Musculoskeletal and connective tissue disorders) | 3
Pain - chest wall (Musculoskeletal and connective tissue disorders) | 7
Pain - headache (Nervous system disorders) | 5
Pain - joint (Musculoskeletal and connective tissue disorders) | 1
Pain - limb (Musculoskeletal and connective tissue disorders) | 3
Pain - liver (Gastrointestinal disorders) | 1
Pain - muscle (Musculoskeletal and connective tissue disorders) | 15
Pain - neuralgia/peripheral nerve (Nervous system disorders) | 1
Pain - pleura (Respiratory, thoracic and mediastinal disorders) | 1
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3
Airway obstruction/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 188
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary/obstruction/stenosis of airway (bronchus) (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/others (Respiratory, thoracic and mediastinal disorders) | 6
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 1
Obstruction/GI (Gastrointestinal disorders) | 4
Renal failure (Renal and urinary disorders) | 10
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intraoperative complications (Surgical and medical procedures) | 1
Antiphospholipid syndrome (Immune system disorders) | 1
Flu-like syndrome (General disorders) | 1
Ill-defined disorder (General disorders) | 1
Syndromes/other-superior cava vein (Injury, poisoning and procedural complications) | 9
Uncoded (General disorders) | 2
Phlebitis (Vascular disorders) | 2
Thrombosis/embolism (Vascular disorders) | 25
Vascular/other (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib 150 mg/Day (N=1797)
Rhinitis (Infections and infestations) | 14
Allergic reaction (Immune system disorders) | 3
Vasculitis (Vascular disorders) | 3
Hearing (Ear and labyrinth disorders) | 5
Tinnitus (Ear and labyrinth disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 89
Platelets (Investigations) | 8
Neutrophils (Investigations) | 7
Leucocytes (Investigations) | 4
Lymphopenia (Investigations) | 1
Band neutrophil percentage increased (Investigations) | 1
Cardiac arrhythmia (Cardiac disorders) | 27
Vasovagal episodes (Nervous system disorders) | 3
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 8
Cardiac ischemia (Cardiac disorders) | 7
Hypotension (Vascular disorders) | 7
Cardiopulmonary arrest (Cardiac disorders) | 6
Hypertension (Vascular disorders) | 5
Left ventricular systolic dysfunction (Cardiac disorders) | 5
Right ventricular dysfunction (Cardiac disorders) | 2
Valvular heart disease (Cardiac disorders) | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Pericarditis (Cardiac disorders) | 1
Asthenia (General disorders) | 650
Fever (General disorders) | 210
Weight loss (Investigations) | 91
Insomnia (Psychiatric disorders) | 67
Constitutional symptoms/other (General disorders) | 42
Sweating (Skin and subcutaneous tissue disorders) | 10
Mucosal dryness (Gastrointestinal disorders) | 6
Pallor (Vascular disorders) | 6
Inflammation (General disorders) | 5
Opioid abuse (Social circumstances) | 3
Rigors/chills (General disorders) | 3
Drug abuser (Social circumstances) | 1
Hypothermia (General disorders) | 1
Weight gain (Investigations) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Rash (Skin and subcutaneous tissue disorders) | 897
Dermatology/skin-other (Skin and subcutaneous tissue disorders) | 307
Acne (Skin and subcutaneous tissue disorders) | 152
Dry skin (Skin and subcutaneous tissue disorders) | 137
Pruritus (Skin and subcutaneous tissue disorders) | 95
Alopecia (Skin and subcutaneous tissue disorders) | 92
Nail changes (Skin and subcutaneous tissue disorders) | 71
Ulceration (Skin and subcutaneous tissue disorders) | 15
Hand foot skin reaction (Skin and subcutaneous tissue disorders) | 9
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 6
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 4
Flushing (Vascular disorders) | 3
Burn (Injury, poisoning and procedural complications) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1
Cushingoid (Endocrine disorders) | 6
ADH (Investigations) | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 631
Anorexia (Metabolism and nutrition disorders) | 462
Vomiting (Gastrointestinal disorders) | 204
Nausea (Gastrointestinal disorders) | 196
Mucositis (Gastrointestinal disorders) | 167
Constipation (Gastrointestinal disorders) | 110
Dysphagia (Gastrointestinal disorders) | 49
Dyspepsia/heartburn (Gastrointestinal disorders) | 40
Xerostomia (Gastrointestinal disorders) | 36
Gastrointestinal/other (Gastrointestinal disorders) | 35
Dysgeusia (Nervous system disorders) | 17
Hemorrhoids (Gastrointestinal disorders) | 8
Incontinence, anal (Gastrointestinal disorders) | 7
Distension (Gastrointestinal disorders) | 6
Flatulence (Gastrointestinal disorders) | 5
Ileus GI (Gastrointestinal disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 4
Esophagitis (Gastrointestinal disorders) | 4
Enteritis (Gastrointestinal disorders) | 2
Intestinal perforation (Gastrointestinal disorders) | 2
Taste Alteration (dysgeusia) (Nervous system disorders) | 1
Anal fistula (Gastrointestinal disorders) | 1
Obstruction/GU (Gastrointestinal disorders) | 1
Tooth disorder (Gastrointestinal disorders) | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 167
Hemorrhage/GI (Gastrointestinal disorders) | 43
Hemorrhage/GU (Renal and urinary disorders) | 14
Petechiae (Skin and subcutaneous tissue disorders) | 6
Hemorrhage/other (General disorders) | 3
Liver dysfunction (Hepatobiliary disorders) | 10
Hepatobiliary/other (Hepatobiliary disorders) | 6
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic cysts (Hepatobiliary disorders) | 1
Infection NOS (Infections and infestations) | 148
Infection - conjunctiva (Infections and infestations) | 108
Infection - lung (pneumonia) (Infections and infestations) | 51
Infection - ungual (nail) (Infections and infestations) | 51
Infection - urinary tract nos (Infections and infestations) | 31
Infection - skin (cellulitis) (Infections and infestations) | 29
Infection - bronchus (Infections and infestations) | 18
Infection - eye nos (Infections and infestations) | 17
Infection - soft tissue nos (Infections and infestations) | 13
Infection - upper aerodigestive nos (Infections and infestations) | 13
Infection - pharynx (Infections and infestations) | 9
Infection - blood (Infections and infestations) | 8
Infection - lip/perioral (Infections and infestations) | 7
Infection - anal/perianal (Infections and infestations) | 5
Infection - upper airway nos (Infections and infestations) | 4
Tooth infection (Infections and infestations) | 4
Infection - vagina (Infections and infestations) | 3
Infection - auditory ear (Infections and infestations) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Gallbladder infection (Infections and infestations) | 2
Infection - brain (encephalitis, infectious) (Infections and infestations) | 2
Infection - sinus (Infections and infestations) | 2
Infection - bone (osteomyelitis) (Infections and infestations) | 1
Infection - kidney (Infections and infestations) | 1
Infection - liver (Infections and infestations) | 1
Infection - salivary gland (Infections and infestations) | 1
Infection - dental-tooth (Infections and infestations) | 1
Infection - peritoneal cavity (Infections and infestations) | 1
Infection - wound (Infections and infestations) | 1
Infection - appendix (Infections and infestations) | 1
Infection - catheter-related (Infections and infestations) | 1
Infection - colon (Infections and infestations) | 1
Infection - vulva (Infections and infestations) | 1
Edema limb (General disorders) | 80
Edema (General disorders) | 33
Edema head and neck (General disorders) | 12
Lymphatic/other (General disorders) | 2
Bilirubin (Investigations) | 23
Hyperglycemia (Metabolism and nutrition disorders) | 17
ALT (Investigations) | 14
AST (Investigations) | 14
Alkaline phosphatase (Investigations) | 11
Hypercalcemia (Metabolism and nutrition disorders) | 11
GGT (Investigations) | 10
Hyperkalemia (Metabolism and nutrition disorders) | 9
Hypocalcemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 7
Metabolic lab/other (Metabolism and nutrition disorders) | 6
Hyperuricemia (Metabolism and nutrition disorders) | 5
Hypercholesterolemia (Investigations) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypoglycemia (Metabolism and nutrition disorders) | 2
Acidosis (Metabolism and nutrition disorders) | 1
Amylase (Investigations) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
CPK (Investigations) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Alkalosis (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Musculoskeletal/other (Musculoskeletal and connective tissue disorders) | 77
Muscle weakness (Musculoskeletal and connective tissue disorders) | 24
Fracture (Injury, poisoning and procedural complications) | 12
Ascites (Gastrointestinal disorders) | 10
Gait (General disorders) | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 6
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Trismus (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 94
Neuropathy/sensory (Nervous system disorders) | 74
Ataxia (Nervous system disorders) | 57
Confusion (Psychiatric disorders) | 55
Neurology/other (Nervous system disorders) | 53
Mood alteration-anxiety (Psychiatric disorders) | 51
Mood alteration-depression (Psychiatric disorders) | 45
Neuropathy/motor (Nervous system disorders) | 38
Somnolence (Nervous system disorders) | 38
Cognitive disturbance (Nervous system disorders) | 28
Speech impairment (Nervous system disorders) | 27
Mood alteration-agitation (Psychiatric disorders) | 23
CNS ischemia (Nervous system disorders) | 16
Tremor (Nervous system disorders) | 16
Syncope (Nervous system disorders) | 15
Seizures (Nervous system disorders) | 15
Mood alteration (Psychiatric disorders) | 14
Memory impairment (Nervous system disorders) | 11
Psychosis (Psychiatric disorders) | 7
Involuntary movement (Nervous system disorders) | 6
Encephalopathy (Nervous system disorders) | 5
Neuropathy cranial (Nervous system disorders) | 5
Mood alteration-depression-anxiety (Psychiatric disorders) | 4
Blurred vision (Eye disorders) | 3
Extrapyramidal disorder (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Eye disorder (Eye disorders) | 48
Watery eye (Eye disorders) | 7
Dry eye (Eye disorders) | 6
Diplopia (Eye disorders) | 5
Keratitis (Eye disorders) | 3
Cataract (Eye disorders) | 2
Vision-flashing lights/floaters (Eye disorders) | 1
Pain nos (General disorders) | 229
Pain - chest wall (Musculoskeletal and connective tissue disorders) | 211
Pain - muscle (Musculoskeletal and connective tissue disorders) | 139
Pain - abdomen nos (Gastrointestinal disorders) | 108
Pain - headache (Nervous system disorders) | 97
Pain - joint (Musculoskeletal and connective tissue disorders) | 95
Pain - bone (Musculoskeletal and connective tissue disorders) | 78
Pain - limb (Musculoskeletal and connective tissue disorders) | 51
Pain - pleura (Respiratory, thoracic and mediastinal disorders) | 25
Pain - neck (Musculoskeletal and connective tissue disorders) | 21
Pain - neuralgia/peripheral nerve (Nervous system disorders) | 18
Pain - liver (Hepatobiliary disorders) | 8
Pain - eye (Eye disorders) | 5
Pain - throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 5
Pain - tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Pain - face (General disorders) | 2
Pain - Kidney (Renal and urinary disorders) | 2
Pain - foot (Musculoskeletal and connective tissue disorders) | 2
Pain - dental/teeth/peridontal (Gastrointestinal disorders) | 1
Pain - ear (Ear and labyrinth disorders) | 1
Pain - rectum (Gastrointestinal disorders) | 1
Pain - scalp (Skin and subcutaneous tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 691
Cough (Respiratory, thoracic and mediastinal disorders) | 436
Pulmonary/other (Respiratory, thoracic and mediastinal disorders) | 138
Voice changes (Respiratory, thoracic and mediastinal disorders) | 87
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 18
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 7
Pulmonary/obstruction/stenosis of airway (bronchus) (Respiratory, thoracic and mediastinal disorders) | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3
Chest tube drainage or leak (Respiratory, thoracic and mediastinal disorders) | 1
Trachael fistula (Respiratory, thoracic and mediastinal disorders) | 1
Airway obstruction/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1
Renal failure (Renal and urinary disorders) | 39
Cystitis (Renal and urinary disorders) | 12
Urinary frequency (Renal and urinary disorders) | 11
Renal/other (Renal and urinary disorders) | 8
Obstruction/GI (Gastrointestinal disorders) | 4
Incontinence, urinary (Renal and urinary disorders) | 2
Urine colour change (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Urogenital disorder (Renal and urinary disorders) | 1
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Sexual/reproductive function (Reproductive system and breast disorders) | 3
Irregular menstruation (Reproductive system and breast disorders) | 2
Vaginal dryness (Reproductive system and breast disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Intraoperative complications (Surgical and medical procedures) | 1
Flu-like syndrome (General disorders) | 102
Syndromes/other-superior cava vein (Injury, poisoning and procedural complications) | 15
Syndromes/other (General disorders) | 3
Antiphospholipid syndrome (Immune system disorders) | 1
Ill-defined disorder (General disorders) | 1
Uncoded (General disorders) | 11
Thrombosis/embolism (Injury, poisoning and procedural complications) | 42
Vascular/other (Vascular disorders) | 10
Phlebitis (Vascular disorders) | 7

LIMITATIONS AND CAVEATS:
Nonserious adverse events presented in this record include all adverse events reported during the study, not just nonserious events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.